CLINICAL TRIAL: NCT05688449
Title: Investigation of the Effect of Epidural Analgesia Combined With General Anesthesia on Burst Suppression Rate in Electroencephalogram Based Anesthesia Management
Brief Title: Effect of Epidural Analgesia on Burst Suppression
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20220609
Record Dates: First submitted 2022-11-07; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Post-operative Delirium; Cognitive Dysfunction; Electroencephalography
Keywords: burst suppression; delirium; electroencephalography; anesthesia; regional anesthesia
MeSH Terms: conditions — Emergence Delirium; Cognitive Dysfunction; Delirium | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epidural analgesia (Active Comparator): Eeg monitoring will be implemented with Sedline monitor(Masimo Irvine CA) 5 minutes before epidural catheter insertion, 30 minutes after epidural catheter insertion, during surgery and 5 minutes after extubation.
  Interventions: Drug: Bupivacaine-fentanyl
- placebo (Placebo Comparator): Eeg monitoring will be implemented with Sedline monitor (Masimo Irvine CA) 5 minutes before epidural catheter insertion, 30 minutes after epidural catheter insertion, during surgery and 5 minutes after extubation.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Bupivacaine-fentanyl — A 20 ml bolus of 2 mcg/ml fentanyl + 0.125% bupivacaine solution will be administered to the bupivacaine group via the epidural catheter, and 5ml/hour infusion will be started.
  Arms: Epidural analgesia
Drug: Saline — A 20 ml bolus of saline will be administered to the saline group via the epidural catheter, and 5ml/hour infusion will be started.
  Arms: placebo

SUMMARY:
It has been shown in previous studies that burst suppression has an effect on the development of postoperative delirium (POD) and postoperative cognitive dysfunction (POCD). With the development of technology, EEG-based anesthesia management is getting more and more attention. In particular, methods that reduce anesthetic drug consumption are expected to prevent POD and POCD by reducing burst suppression. There are studies that show that epidural analgesia applications reduce general anesthesia drug consumption in patients receiving general anesthesia. In this study, investigators want to investigate the effect of epidural analgesia combined with general anesthesia on burst suppression. POD and POCD development in these patients will be examined as secondary objectives.

DETAILED DESCRIPTION:
Postoperative delirium (POD) is an acute cognitive disorder characterized by inattention, disorganized thinking, and a fluctuating course that develops over hours or days. Although delirium depends on the type of surgery, it is a common postoperative complication with an incidence of 10%-70%. POD causes an increase in mortality, morbidity and health care costs. Risk factors for POD; age, type and duration of surgery, inadequate pain control, type of anesthesia, anemia, transfusion, and preoperative cognitive impairment. In recent years, it has been emphasized that POD can be reduced with the widespread use of electroencephalogram (EEG) based anesthesia management and optimization of anesthetic drugs according to EEG patterns. EEG consists of 6 waveforms: slow, delta, theta, alpha, beta and gamma. Behavioral and neurophysiological patterns caused by anesthetic drugs are associated with different electroencephalogram waveforms. Recent developments in the introduction of EEG-based monitors have made significant contributions to the understanding of the fundamental changes in brain activity caused by anesthetic agents. Today, there are EEG-based anesthesia depth monitors such as bispectral index (BIS) (Medtronic, USA) or Sedline (Masimo Irvine CA). These monitors make it easier to optimize the depth of anesthesia with the numerical data obtained as a result of some calculations as well as the raw EEG. The burst suppression (BS) pattern on the EEG shows a decrease in brain neuronal activity and metabolic activity. Burst suppression can be induced by anesthetic drugs that modulate γ-aminobutyric acid type A receptors. Although sometimes deliberately induced for therapeutic purposes to treat refractory status epilepticus or increased intracranial pressure, burst suppression is generally considered potentially harmful and should be avoided.Studies conducted in recent years have shown the relationship between intraoperative burst suppression (BS) and POD. POD; It can be reduced by continuous EEG monitoring, reducing the dose of propofol, preferring regional anesthesia, effective postoperative pain control, early mobilization, and early postoperative discharge. Interventions that can reduce the development of postoperative delirium will be important for public health. Epidural analgesia can be used effectively in perioperative analgesia. It has been reported in the literature that epidural analgesia combined with general anesthesia reduces the amount of hypnotic drug required to achieve similar depth of anesthesia compared to general anesthesia alone. There is no study in the literature on whether the combination of epidural analgesia and general anesthesia reduces BS in EEG-based anesthesia applications. Our primary aim in this study is to evaluate whether the combination of general anesthesia and epidural analgesia reduces BS in EEG-based anesthesia in patients undergoing total hip and knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Physical Status 1-3
* Hip or knee arthroplasty surgery

Exclusion Criteria:

* severe renal failure (need for renal replacement therapy)
* severe liver failure (child-pudg grade c)
* body mass index >40
* long-term use of some drugs (sedatives, tricyclic antidepressants, narcotic painkillers)
* having a disease related to the nervous system
* having a psychiatric disease
* having a history of substance abuse
* having consumed 2 or more glasses of alcohol per day in the last 1 year
* contraindications for neuraxial block
* allergy to drugs to be used
* emergency surgeries
* patient's refusal to accept the procedure
* hearing and visual impairment
* anesthesia awareness history
* preoperative delirium

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-07-30 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
burst suppression | Form beginning of anesthesia induction to the end of anesthesia(During perioperative period)
  burst suppression rate

SECONDARY OUTCOMES:
postoperative two days delirium rate | Within the first two postoperative days
  Screening of the patients regarding a postoperative delirum by Confusion Assessment Method for the ICU.
Postoperative cognitive dysfunction rate | Participants will be called for control in the postoperative 1st and 3rd months.
  Screening of the patients regarding a postoperative cognitive dysfunction by the telephone Montreal Cognitive Assessment(t-MoCA)

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University Hospital, Istanbul, Fatih, Turkey (Türkiye)